CLINICAL TRIAL: NCT03445429
Title: 3D- vs. 4K-display System - Influence of "State-of-the-art"-Display Technique on Surgical Performance
Brief Title: Influence of 3D- vs. 4K-display System on Surgical Performance
Acronym: IDOSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Principal Investigator, Roger Wahba, MD, PhD, Priv.-Doz. Dr. med. Roger Wahba, Universitätsklinikum Köln
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 17-388
Record Dates: First submitted 2018-02-07; First posted 2018-02-26 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Surgical Performance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-display system (Experimental): Subjects in this arm will perform the tasks on the minimal-invasive training set-up first with the 3D-display system. Then they will do the NASA task load index questionnaire. After that they will perform the tasks with the 4 K-display system. After that again a NASA Task load index questionnaire is performed.
  Interventions: Other: 3D-display system
- 4K-display system (Experimental): Subjects in this arm will perform the tasks on the minimal-invasive training set-up first with the 4K-display system. Then they will do the NASA task load index questionnaire. After that they will perform the tasks with the 3D-display system. After that again a NASA Task load index questionnaire is performed.
  Interventions: Other: 4K-display system

INTERVENTIONS:
Other: 3D-display system — The subjects will perform tasks on a minimal-invasive/laparoscopic training set-up. They will perform the tasks with a 3D-display system or a 4K-display system. The intervention type 3D-display system means that the training-set up is performed first with 3D-display system an after that with the 4K-display system.
  Arms: 3D-display system
Other: 4K-display system — The subjects will perform tasks on a minimal-invasive/laparoscopic training set-up. They will perform the tasks with a 3D-display system or a 4K-display system. The intervention type 4K-display system means that the training-set up is performed first with 4K-display system and after that with the 3D-display system.
  Arms: 4K-display system

SUMMARY:
Modern display technique seems to optimize visualization in minimal-invasive surgery. Many systems are available right now with a fundamental difference between the passive polarizing 3-dimensional (3D) and 2-dimensional (2D) technique. Data seems to show a benefit for the 3D technique in the visualization of the operative field. This could lead to more precision in minimal-invasive surgery. 2D-systems with high resolution of 4.096 x 2.180 pixels (4K) could be a promising alternative. This study wants to evaluate if 3D- or 4K- display technique could optimize surgeons´ view and improve the performance during minimal-invasive surgery. Therefore medical students and surgeons of different experience levels will perform surgical tasks on a minimal-invasive training system.They will be randomized to use first the 3D- or the 4K-display system in the training set-up. After completing the tasks with one system the minimal-invasive training set-up will be repeated with the other display system. NASA (National Aeronautics and Space Administration) task load index is evaluated after each round. The ability for stereoscopic vision is tested after finishing the complete training set-up with both systems. The primary outcome parameter surgical performance will be evaluated in this study defined as the performance time and the number of defined mistakes made during each task.

ELIGIBILITY:
Inclusion Criteria:

* medical student
* medical doctor
* informed consent signed

Exclusion Criteria:

* known deficit of stereoscopic view
* experience with the tasks of the minimal-invasive training set-up
* not able to use both hands for minimal-invasive training set-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Surgical Performance Time | immediately after tasks are performed, Day 1
  The surgical performance time is defined as time needed to complete the tasks at the minimal-invasive trainer. the time is measured in seconds
Surgical Performance Errors | immediately after tasks are performed, Day 1
  it is measured once directly after completing the task with the 3D performance time and the number of errors: the surgical performance errors are defined as the number of defined errors made during the performance of the tasks at the minimal invasive trainer surgical performance errors = number of errors

SECONDARY OUTCOMES:
Task Load | immediately after tasks are performed, Day 1
  task load felt by the subjects evaluated by NASA task load index, after tasks with 3 D- and 4 K- systems are completed NASA task load index is evaluated once
Learning curve | immediately after tasks with both systems (3D and 4K) are performed, Day 1
  Learning curve after the completeness of the tasks
Stereoscopic view Bagolini | immediately after tasks with both systems (3D and 4K) are performed, Day 1
  Qualitative test for assesment of stereoscopic view units : positive /negative/diplopia
Stereoscopic view Lang I/II | immediately after tasks with both systems (3D and 4K) are performed, Day 1
  Semi-quantitative test for assesment of stereoscopic view units : arc seconds
Stereoscopic view Titmus | immediately after tasks with both systems (3D and 4K) are performed, Day 1
  Semi-quantitative test for assesment of stereoscopic view units : arc seconds (fly at 3550 arc seconds, animals at 400, 200, 100 arc seconds,rings at 800, 400, 200, 140, 100, 80, 60, 50, 40 arc seconds)
Stereoscopic view TNO | immediately after tasks with both systems (3D and 4K) are performed, Day 1
  Semi-quantitative test for assesment of stereoscopic view units: arc seconds (480, 240, 120, 60, 30, 15)
Stereoscopic view Cover | immediately after tasks with both systems (3D and 4K) are performed, Day 1
  qualitative test for assesment of stereoscopic view units: phoria/tropia

CONTACTS AND LOCATIONS:
Overall Officials: Roger Wahba, MD, PhD, Principal Investigator — Universitätsklinikum Köln
Locations (1):
- University of Cologne, Department of General, Visceral and Cancer Surgery, Cologne, Germany

REFERENCES:
- [Derived] Gietzelt C, Datta R, Busshoff J, Bruns T, Wahba R, Hedergott A. The influence of stereoscopic vision on surgical performance in minimal invasive surgery-a substudy of the IDOSP-Study (Influence of 3D- vs. 4 K-Display Systems on Surgical Performance in minimal invasive surgery). Langenbecks Arch Surg. 2022 Nov;407(7):3069-3078. doi: 10.1007/s00423-022-02608-3. Epub 2022 Jul 22. PMID 35869334
- [Derived] Wahba R, Datta RR, Hedergott A, Busshoff J, Bruns T, Kleinert R, Dieplinger G, Fuchs H, Gietzelt C, Moller D, Hellmich M, Bruns CJ, Stippel DL. 3D vs. 4K Display System - Influence of "State-of-the-art"-Display Technique On Surgical Performance (IDOSP-Study) in minimally invasive surgery: protocol for a randomized cross-over trial. Trials. 2019 May 28;20(1):299. doi: 10.1186/s13063-019-3330-7. PMID 31138290